CLINICAL TRIAL: NCT00253019
Title: A Comparison of Continuation Rates for Three Hormonal Contraceptive Methods (Oral Contraceptive Pills, Depo Provera and Ortho Evra) Among Women Seeking First Trimester Abortion.
Brief Title: A Comparison of Continuation Rates for Three Hormonal Contraceptive Methods
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Carrie Cwiak, Principal Investigator, Emory University
Other Study IDs: 518-2003
Record Dates: First submitted 2005-11-14; First posted 2005-11-15 (Estimated); Results first posted 2013-08-09 (Estimated); Last update posted 2013-08-21 (Estimated); Status verified 2013-08

CONDITIONS: Contraception
Keywords: birth control; continuation; abortion; contraception

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will assess the continuation rates among women using oral contraceptive pills, Depo-Provera and Ortho Evra following a first trimester abortion.

DETAILED DESCRIPTION:
Unintended pregnancy rates among women in the United States continue to surpass that of the rest of the developed world at great cost to society. Contraceptive failure has been attributed to poor compliance with contraceptive methods and results in unintended pregnancies. This study will evaluate the 3-month continuation rates among women using the oral contraceptive pill and Depo-Provera. It will also assess the continuation rates of Ortho Evra®, which has not previously been studied in the adolescent population. This study will provide information with regard to pregnancy rates and 3-month patterns of use of contraception among women seeking first-trimester abortion. It will also assess other factors contributing to successful contraception such as the use of emergency contraception and concomitant condom use. The results of this study will be used to inform the practice of providers who provide reproductive health care to women and add to the sparse body of literature available comparing the success of different contraceptive methods used by women.

ELIGIBILITY:
Inclusion Criteria:

* Age 13-45 women presenting at the ambulatory surgery at Grady Memorial Hospital who want to use either oral contraceptive pills, ortho evra or depo provera?

Exclusion Criteria:

* Leaving the Atlanta area within 6 months?
* Desires pregnancy within the next 6 months?
* Unable to provide contact information?
* Contraindications to hormonal contraceptive?

Ages: 13 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Participants were recruited from a indigent, urban, African American population.
Sampling Method: Non-Probability Sample
Enrollment: 321 (Actual)
Dates: Start 2004-10; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carrie Cwiak, MD, MPH, Principal Investigator — Emory University
Locations (1):
- Grady Memorial Hospital, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from a medical clinic beginning in 10/2004 through 11/2005.
Pre-assignment Details: All patients were invited to participate.
Groups:
- Oral Contraceptive: Participants self-selected to receive oral contraceptives.
- Depo Provera: Participants self-selected to receive Depo Provera
- Ortho Evra: Participants self-selected to receive Ortho Evra.
Period: Overall Study
Arm/Group | Oral Contraceptive | Depo Provera | Ortho Evra
Started | 111 | 109 | 101
Completed | 82 | 78 | 83
Not Completed | 29 | 31 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Contraceptive | Depo Provera | Ortho Evra | Total
Number analyzed (Participants) | 111 | 109 | 101 | 321
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 111 | 109 | 101 | 321
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 111 | 109 | 101 | 321
  Male | 0 | 0 | 0 | 0
The measure is of what contraceptive method the participants chose to use [Number; unit: participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 111 | 109 | 101 | 321
  >=65 years | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Continuation Rates
Description: We followed subjects to evaluate the continuation rates for subjects receiving oral contraceptive pills, Depo Provera and Ortho Evra.
Time Frame: 3 months
Population: It was a convenience sample.
Measure: Number; unit: participants
Arm/Group | Oral Contraceptive | Depo Provera | Ortho Evra
Number analyzed (Participants) | 111 | 109 | 101
participants | 82 | 78 | 83

ADVERSE EVENTS:
Groups:
- Oral Contraceptives: participants self-selected to take oral contraceptives
- Depo Provera: Participants self-selected to use depo provera
Arm/Group | Oral Contraceptives | Depo Provera | Ortho Evra
Serious Adverse Events (participants affected / at risk) | 0/111 | 0/109 | 0/101
Other Adverse Events (participants affected / at risk) | 0/111 | 0/109 | 0/101

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes